CLINICAL TRIAL: NCT00441844
Title: Phase 2 Study Examining the Effect of Simvastatin vs Placebo on Monocyte Function and Inflammation in Patients With Type 1 Diabetes
Brief Title: Monocyte Function and Inflammation in Type 1 Diabetes and Its Modulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDFT1DMSIMVA; UCD IRB # 200210057
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Type 1 Diabetes
Keywords: diabetes, statin, monocyte, crp, inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
Type I diabetes (T1DM) is associated with an increased risk of vascular complications. While the precise mechanism(s) by which diabetes accelerates atherosclerosis has not been elucidated, several lines of evidence point to the role of increased inflammation in the pathogenesis of these vasculopathies. The monocyte-macrophage is a pivotal cell in atherogenesis and is readily accessible for study. However, there is scanty data on monocyte function and inflammation in T1DM. Simvastatin, a HMG-CoA reductase inhibitor, has recently been shown to reduce cardiovascular events in diabetic patients (T1DM and T2DM in the Heart Protection Study). Recent studies demonstrate that simvastatin decreased C-reactive protein and decreased pro-atherogenic activity of monocytes in non-diabetic subjects. However, there is a paucity of data on the effect of simvastatin on inflammation and monocyte function in Type 1 diabetes.

Thus, the purpose of this study is Aim 1) to assess biomarkers of inflammation in T1DM compared to matched controls (n=50/group). Aim 2) Also, we will assess the effect of simvastatin (20mg/day) therapy on inflammation and monocyte function in T1DM in a randomized, placebo-controlled, double blind trial.

DETAILED DESCRIPTION:
Type I diabetes (T1DM) is associated with an increased risk of vascular complications. While the precise mechanism(s) by which diabetes accelerates atherosclerosis has not been elucidated, several lines of evidence point to the role of increased inflammation in the pathogenesis of these vasculopathies. The monocyte-macrophage is a pivotal cell in atherogenesis and is readily accessible for study. However, there is scanty data on monocyte function and inflammation in T1DM. Simvastatin, a HMG-CoA reductase inhibitor, has recently been shown to reduce cardiovascular events in diabetic patients (T1DM and T2DM in the Heart Protection Study). Recent studies demonstrate that simvastatin decreased C-reactive protein and decreased pro-atherogenic activity of monocytes in non-diabetic subjects. However, there is a paucity of data on the effect of simvastatin on inflammation and monocyte function in Type 1 diabetes.

Thus, the purpose of this study is Aim 1) to assess biomarkers of inflammation in T1DM compared to matched controls (n=50/group). Aim 2) Also, we will assess the effect of simvastatin (20mg/day) therapy on inflammation and monocyte function in T1DM in a randomized, placebo-controlled, double blind trial.

At baseline and post-therapy, fasting blood will be obtained for routine laboratories (including lipid profile, glucose, glycated hemoglobin), free fatty acid levels, biomarkers of inflammation [high sensitive C-reactive protein, plasma soluble cell adhesion molecules (sVCAM,sICAM, sE-selectin and sP-selectin) , CD40 ligand, monocyte pro-atherogenic activity (superoxide anion, monocyte chemotactic protein-1, interleukin (IL)-1b, IL-6 and tumor necrosis factor-a release, adhesion to human aortic endothelium, CD40 expression)] etc., and 24-hour urine for microalbumin

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetic patients (onset < 20years and on insulin therapy since diagnosis) without clinical macrovascular complications, present age > 20 years with duration of diabetes > 1yr.

Exclusion Criteria:

* HbA1c over the last year >10%
* Patients on glucophage and/or the thiazolidenediones will be excluded, since these drugs appear to be anti-inflammatory.
* Theumatoid arthritis;
* Abnormal liver function,
* Hypo- or hyperthyroidism;
* Malabsorption;
* Steroid therapy,
* Anti-inflammatory drugs except aspirin (81mg/day)
* Pregnancy,
* Lactation,
* Smoking,
* Abnormal complete blood count; and
* Alcohol consumption > 1 oz/day

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-10; Study Completion 2005-07

PRIMARY OUTCOMES:
HsCRP
Monocyte function

SECONDARY OUTCOMES:
Plasma biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Ishwarlal Jialal', MD, PhD, Principal Investigator — UCDavis Professor
Locations (1):
- UCDavis Medical Center, Sacramento, California, United States